CLINICAL TRIAL: NCT03490903
Title: Coronary Angiography THerapeutic Virtual Reality: Investigating the Effect of Virtual Reality on Procedural Anxiety, Pain and Vasospasm
Brief Title: Coronary Angiography THerapeutic Virtual Reality
Acronym: CATH-VR
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No patients enrolled
Sponsor: University of California, Los Angeles (Other)
Collaborators: AppliedVR Inc. (Industry)
Responsible Party: Principal Investigator, David J. Cho, MD, MBA, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB#18-000026
Record Dates: First submitted 2018-03-30; First posted 2018-04-06 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Virtual Reality; Atherosclerosis; Coronary Artery Disease; Anxiety; Pain, Acute; Vasospasm;Peripheral
Keywords: virtual reality; anxiety; vasospasm; pain; coronary artery angiography; angiogram; VR
MeSH Terms: conditions — Atherosclerosis; Coronary Artery Disease; Anxiety Disorders; Acute Pain; Pain | interventions — Fentanyl; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VR with or without Moderate Sedation (Experimental): Patients randomized to receive a Virtual Reality Intervention will be fitted with a VR headset and headphones and undergo a continuous immersive meditation experience. This will begin immediately prior to the start of the procedure, and continue until the procedure is completed.
  Patient pain and anxiety levels will be frequently assessed by procedure operator and circulating nurse, and pain medication or anxiolytic medications will be administered in the absence of contraindications. Baseline amounts of sedation pre-procedurally will not be used in either arm. Pain and Anxiety Scores will be assessed pre, intra, and post-procedurally. If no contraindications, the operator will decide upon how much sedation medication to administer if indicated or requested. This is the usual manner in which pain and anxiety is treated in the cath lab.
  Interventions: Device: Virtual Reality; Drug: Fentanyl Injection; Drug: Midazolam injection
- Moderate Sedation without VR (Active Comparator): Subjects randomized to the comparison arm will not undergo the Virtual Reality Intervention. Baseline amounts of sedation pre-procedurally will not be used in either arm. Subjects will be assessed periodically by physicians and/or circulating nurses for their pain and anxiety levels. The patient may also prompt the staff that they are anxious or in pain, and if no contraindications, the operator will decide upon how much medication to administer. This is the usual manner in which pain and anxiety is treated in the cath lab.
  Interventions: Drug: Fentanyl Injection; Drug: Midazolam injection

INTERVENTIONS:
Device: Virtual Reality — Subjects undergoing the Virtual Reality Intervention will be fitted with a VR headset and headphones, and undergo an immersive meditation experience provided by AppliedVR, Inc. The headphones will not be noise-cancelling, and the subject will be able to communicate with the physician or circulating nurse if needed.
  Arms: VR with or without Moderate Sedation
Drug: Fentanyl Injection — Fentanyl is commonly administered to treat pain during invasive procedures such as coronary angiography. Intravenous fentanyl injection dosages are determined by the physician operator, and administered by the circulating nurse.
Drug: Midazolam injection — Midazolam is commonly administered to treat anxiety during invasive procedures such as coronary angiography. Intravenous midazolam injection dosages are determined by the physician operator, and administered by the circulating nurse.

SUMMARY:
The CATH-VR study will investigate the effect of virtual reality (VR) on patient pain, anxiety, and radial artery vasospasm during coronary angiography. Our hypothesis is that the use of VR will decrease patient anxiety and pain via validated scoring systems, as well as show a low rate of vasospasm of the radial artery. In addition, we hypothesize that the amount of opioid and benzodiazepine medications utilized for procedural sedation will be lower in the intervention arm. VR has gained recent attraction as an alternative or adjunctive treatment option for pain, but its effect on reducing procedural sedation has not been studied. We propose a single center, randomized control pilot study to further investigate. The patient population will include adults older than 18 years who present for outpatient diagnostic coronary angiography.

DETAILED DESCRIPTION:
We plan to conduct a prospective, unblinded, randomized control pilot study to test our hypothesis that the use of VR will decrease patient anxiety and pain via validated scoring systems, as well as show a low rate of vasospasm of the radial artery.

Patients will be eligible if they are greater than 18 years of age and undergoing an elective outpatient coronary angiogram with or without percutaneous intervention. Exclusion criteria will include patients with claustrophobia, seizure disorder, motion sickness, stroke within the past year, dementia, nausea, isolation status for infection control or those who do not wish to participate.

Outpatients undergoing routine coronary angiography with or without possible percutaneous intervention will be screened for enrollment criteria. Those who agree to participate will be randomized to either the intervention or control arm. Those randomized to the intervention arm and agree to participate in the study will wear a VR Headset and headphones; those who are randomized to the control will receive the standard of care, which is moderate sedation for patient anxiolysis and pain control during the case. In both arms, the patient and operator will still be able to communicate verbally if needed to assess for pain, to ask questions, or to ask for anxiolytic or analgesic medications as needed. The procedure will be completed when vascular sheaths are just about to be removed.

ELIGIBILITY:
Inclusion Criteria:

- Age greater than or equal to 18 years undergoing diagnostic coronary angiogram

Exclusion Criteria:

* Claustrophobia
* Seizure disorder
* Motion sickness
* Stroke within the past year
* Dementia
* Nausea
* Isolation status for infection control
* Do not wish to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-06-01 (Estimated); Primary Completion 2018-06-30 (Estimated); Study Completion 2018-06-30 (Estimated)

PRIMARY OUTCOMES:
Radial Artery Vasospasm | Day 1
  Presence or Absence of Radial Artery Vasospasm, determined by procedure operator
Pain | Day 1
  Participants will verbalize their level of pain using the Wong-Baker FACES® Score (0 - 10 point scale, 10 points = worst pain, 0 = no pain).
Anxiety | Day 1
  Participants will verbalize their level of anxiety by using the abbreviated State-Trait Anxiety Inventory 6 Score (Score Range 20-80, higher numbers correlate with higher levels of anxiety in a certain moment)

SECONDARY OUTCOMES:
Total fentanyl sedation | Day 1
  The total dose of fentanyl administered during the procedure
Total midazolam sedation | Day 1
  The total dose of midazolam administered during the procedure

CONTACTS AND LOCATIONS:
Overall Officials: David Cho, MD, Principal Investigator — University of California, Los Angeles

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tashjian VC, Mosadeghi S, Howard AR, Lopez M, Dupuy T, Reid M, Martinez B, Ahmed S, Dailey F, Robbins K, Rosen B, Fuller G, Danovitch I, IsHak W, Spiegel B. Virtual Reality for Management of Pain in Hospitalized Patients: Results of a Controlled Trial. JMIR Ment Health. 2017 Mar 29;4(1):e9. doi: 10.2196/mental.7387. PMID 28356241
- [Background] Gold JI, Mahrer NE. Is Virtual Reality Ready for Prime Time in the Medical Space? A Randomized Control Trial of Pediatric Virtual Reality for Acute Procedural Pain Management. J Pediatr Psychol. 2018 Apr 1;43(3):266-275. doi: 10.1093/jpepsy/jsx129. PMID 29053848
- [Background] Buffum MD, Sasso C, Sands LP, Lanier E, Yellen M, Hayes A. A music intervention to reduce anxiety before vascular angiography procedures. J Vasc Nurs. 2006 Sep;24(3):68-73; quiz 74. doi: 10.1016/j.jvn.2006.04.001. PMID 16952777